CLINICAL TRIAL: NCT02484781
Title: Gait Analyses After Resurfacing Hip Arthroplasty Versus Metal on Metal Total Hip
Brief Title: Gait Analyses After Resurfacing Hip Arthroplasty Versus Metal on Metal Total Hip Arthroplasty, an Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: RMC Groot Klimmendaal (Unknown)
Responsible Party: Principal Investigator, Job van Susante, Dr. JLC van Susante, Rijnstate Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LTC 2015-0576
Record Dates: First submitted 2015-06-09; First posted 2015-06-30 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Difficulty Walking; Gait, Stumbling
Keywords: Gait disorder; Resurfacing Hip Arthroplasty; Total Hip Arthroplasty
MeSH Terms: conditions — Mobility Limitation; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Hip Arthroplasty (Active Comparator): Gait analysis on a trendmill of patients with a well functioning total hip arthroplasty on a trendmill
  Interventions: Other: Gait analysis on a trendmill
- Resurfacing Hip Arthroplasty (Active Comparator): Gait analysis on a trendmill of patients with a well functioning resurfacing hip arthroplasty on a trendmill
  Interventions: Other: Gait analysis on a trendmill

INTERVENTIONS:
Other: Gait analysis on a trendmill — Gait analysis on a trendmill "GRAIL" to analyse spatio-temporal kinetics and kinematics when flat walking and inclining
  Other Names: Gait realtime analysis interactive lab: MOTEK Medical

SUMMARY:
Total hip replacement surgery is a very successful operation with good long-term results. Hip resurfacing arthroplasty is offered as a treatment option for young and active patients with osteoarthritis of the hip. It has been proposed as a treatment option for younger patients because of claims that it preserves femoral bone stock and has better functional outcomes. The assessment of gait after hip replacement surgery may be able to determine functional differences between patients who have undergone total hip replacement / arthroplasty (THA) versus hip resurfacing.

DETAILED DESCRIPTION:
A group of 58 patients, part of a ungoing randomized trial comparing resurfacing hip arthroplasty to metal-on-metal total hip arthroplasty, will be invited to a single gait analysis on a trendmill. All patients have reached a follow up of five years. Patient 's gait will be assessed during two walking sessions, in both sessions spatio-temporal, kinetic and kinematic parameters will be recorded.

* At first when flat walking with increasing speeds to their top walking speed.
* Secondly: when walking at a fixed speed with an increasing incline to their top walking incline.

ELIGIBILITY:
Inclusion Criteria:

* Patient part of randomised controlled trial (RCT) of hip resurfacing versus MoM total hip arthroplasty for symptomatic osteoarthritis of the hip
* Patient must be able to consent to the study (written informed consent)
* Patients who are functioning well post-operatively and not under routine follow up
* Patients who are able to walk without any safety rail assistance on the treadmill

Exclusion Criteria:

* Patient not originally randomised during an RCT of hip resurfacing versus MoM total hip arthroplasty
* Patients who suffer from any neurological or musculoskeletal conditions that might make a gait test dangerous.
* Patients whose cognitive function prevents them from understanding the study
* Patients who have had or are awaiting revision surgery for their hip

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Top walking speed | 5 years postoperative
  Mean top walking speed in kilometers / hour assessed on a trendmill
Walking cadence | 5 years postoperative
  Mean steps / minute at top walking speed assessed on a trendmill
Step length | 5 years postoperative
  Mean step distance in meters at top walking speed assessed on a trendmill
Maximum Push off force (N/kg) per cycle | 5 years postoperative
  Mean ground reaction forces in Newton / kilogram on a trendmill
Maximum weight acceptance (N/kg) per cycle | 5 years postoperative
  Mean ground reaction forces assessed on a trendmill
Mid-stance force (N/kg) per cycle | 5 years postoperative
  Mean ground reaction forces assessed on a trendmill
Hip maximum flexion/extension per cycle | 5 years postoperative
  Mean hip kinematics in degrees assessed on a trendmill
Hip maximum internal/external rotation per cycle | 5 years postoperative
  Mean hip kinematics in degrees assessed on a trendmill

SECONDARY OUTCOMES:
Postoperative hip functionality after hip arthroplasty. | 5 years postoperative
  Postoperative hip function according the Harris Hip Score and Western Ontario and McMaster Universities Osteoarthritis Index
General Health according EurQol-5D | 5 years postoperative
  Health outcome on the EQ-5D questionairre
Physical activity level according the UCLA-activity score | 5 years postoperative
  The University of California at Los Angeles (UCLA) activity score

CONTACTS AND LOCATIONS:
Overall Officials: Job LC Susante, Dr, Principal Investigator — Rijnstate Hospital, orthopedic surgeon
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Background] Aqil A, Drabu R, Bergmann JH, Masjedi M, Manning V, Andrews B, Muirhead-Allwood SK, Cobb JP. The gait of patients with one resurfacing and one replacement hip: a single blinded controlled study. Int Orthop. 2013 May;37(5):795-801. doi: 10.1007/s00264-013-1819-3. Epub 2013 Feb 27. PMID 23443980